CLINICAL TRIAL: NCT02956629
Title: A Phase 2, Open-Label Clinical Trial to Study the Efficacy and Safety of 12 Weeks of the Combination Regimen of MK-3682 + Ruzasvir in Subjects With Chronic Hepatitis C Virus (HCV) Genotype 1, 2, 3, 4, 5 or 6 Infection
Brief Title: Efficacy and Safety of Uprifosbuvir (MK-3682) + Ruzasvir (MK-8408) in Treating Hepatitis C Virus Infection Genotypes 1-6 (MK-3682-041)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated based on review of Phase 2 efficacy data
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3682-041; 2016-003227-37 (EudraCT Number); MK-3682-041 (Other: Merck Protocol Number)
Record Dates: First submitted 2016-11-02; First posted 2016-11-07 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — uprifosbuvir; ruzasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- HCV GT1 (Experimental): Male and female participants with HCV GT1a or GT1b infection take uprifosbuvir 450 mg + RZR 180 mg for 12 weeks.
  Interventions: Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: Ribavirin
- HCV GT2 (Experimental): Male and female participants with HCV GT2 infection take uprifosbuvir 450 mg + RZR 180 mg for 12 weeks.
  Interventions: Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: Ribavirin
- HCV GT3 (Experimental): Male and female participants with HCV GT3 infection take uprifosbuvir 450 mg + RZR 180 mg for 12 weeks.
  Interventions: Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: Ribavirin
- HCV GT4 (Experimental): Male and female participants with HCV GT4 infection take uprifosbuvir 450 mg + RZR 180 mg for 12 weeks.
  Interventions: Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: Ribavirin
- HCV GT5 (Experimental): Male and female participants with HCV GT5 infection take uprifosbuvir 450 mg + RZR 180 mg for 12 weeks.
  Interventions: Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: Ribavirin
- HCV GT6 (Experimental): Male and female participants with HCV GT6 infection take uprifosbuvir 450 mg + RZR 180 mg for 12 weeks.
  Interventions: Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Uprifosbuvir — Participants take 3 tablets each containing 150 mg uprifosbuvir q.d. by mouth.
  Other Names: MK-3682
Drug: Ruzasvir — Participants take 3 capsules each containing 60 mg RZR q.d. by mouth.
  Other Names: MK-8408
Drug: Ribavirin — RBV 200 mg capsules will be taken according to package instructions for a maximum of 16 weeks for any GT that meets virologic futility rules on uprifosbuvir + RZR alone.

SUMMARY:
This is a nonrandomized, multi-site, open-label trial to evaluate a novel two-drug combination regimen (uprifosbuvir [MK-3682] 450 mg + ruzasvir [RZR; MK-8408] 180 mg once daily [q.d.] for 12 weeks) in male and female treatment-naïve (TN) or treatment-experienced (TE) participants with chronic hepatitis C virus (HCV) infection genotype (GT) GT1, GT2, GT3, GT4, GT5, or GT6 who have not previously received HCV direct-acting antiviral (DAA) therapy. Cirrhotic (C) and non-cirrhotic (NC) participants with and without human immunodeficiency virus (HIV) co-infection will be enrolled.

DETAILED DESCRIPTION:
Any GT that meets virologic futility criteria will be given the option of extending treatment with uprifosbuvir + RZR to 16 weeks with ribavirin (RBV) added.

ELIGIBILITY:
Inclusion Criteria:

* has HCV ribonucleic acid (RNA) (≥10,000 IU/mL in peripheral blood) at the time of screening
* has documented chronic HCV GT1, GT2, GT3, GT4, GT5, or GT6 (with no evidence of non-typeable or mixed GT)
* is a female who is not of reproductive potential, or is a female of reproductive potential who agrees to avoid becoming pregnant from two weeks prior to Day 1 through 14 days after the last dose of study drug via abstinence or use of two approved contraceptives
* is C or NC
* if coinfected with HIV, has documented HIV infection prior to Day 1, and either does not use an antiretroviral therapy (ART) or has well-controlled HIV on stable ART (at least 4 weeks prior to study entry)

Exclusion Criteria:

* has evidence of decompensated liver disease
* is C and is Child-Pugh Class B or C, or has a Child-Tucotte-Pugh score >6
* is coinfected with hepatitis B virus (hepatitis B surface antigen or hepatitis B core antibody positive)
* is coinfected with HIV and has a recent (within 6 months prior to screening) opportunistic infection
* has a history of malignancy other than adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or carcinoma in situ within 5 years of signing informed consent
* is C and has evidence (liver imaging within 6 months prior to Day 1) of hepatocellular carcinoma (HCC) or is under evaluation for HCC
* has participated in another investigational drug study within 30 days of signing informed consent
* is a female who is pregnant or breastfeeding or expecting to conceive or donate eggs from Day 1 through 6 months after the last dose of study drug or longer if dictated by local regulations, or is a male who is expecting to donate sperm from Day 1 through 14 days after the last dose of study drug or longer if dictated by local regulations, or is a male whose female partner(s) is/are pregnant or breastfeeding
* has clinically relevant alcohol or drug abuse within 12 months of screening
* has any of the following conditions: organ transplants other than cornea and hair; poor venous access; history of gastric surgery; clinically significant cardiac abnormality/dysfunction; any major medical condition which, in the opinion of the investigator, might interfere with participation; hospitalization within 3 months prior to enrollment; any condition that might require hospitalization; any condition requiring or likely to require chronic systemic administration of corticosteroids, tumor necrosis factor (TNF) antagonists, or immunosuppressant drugs; a life-threatening SAE during screening; or hepatitis not caused by HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lawitz E, Gane E, Feld JJ, Buti M, Foster GR, Rabinovitz M, Burnevich E, Katchman H, Tomasiewicz K, Lahser F, Jackson B, Shaughnessy M, Klopfer S, Yeh WW, Robertson MN, Hanna GJ, Barr E, Platt HL; C-BREEZE-2 Study Investigators. Efficacy and safety of a two-drug direct-acting antiviral agent regimen ruzasvir 180 mg and uprifosbuvir 450 mg for 12 weeks in adults with chronic hepatitis C virus genotype 1, 2, 3, 4, 5 or 6. J Viral Hepat. 2019 Sep;26(9):1127-1138. doi: 10.1111/jvh.13132. Epub 2019 Jul 11. PMID 31108015

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males and females of at least 18 years of age, with chronic Hepatitis C Virus (HCV) infection were enrolled in this study.
Groups:
- HCV Genotype (GT) 1: Male and female participants with HCV GT1a or GT1b infection take uprifosbuvir 450 mg + Ruzasvir (RZR) 180 mg for 12 weeks.
Period: Overall Study
Arm/Group | HCV Genotype (GT) 1 | HCV GT2 | HCV GT3 | HCV GT4 | HCV GT5 | HCV GT6
Started | 78 | 47 | 61 | 56 | 18 | 22
Completed | 73 | 41 | 57 | 55 | 18 | 21
Not Completed | 5 | 6 | 4 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 5 | 3 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HCV GT1 | HCV GT2 | HCV GT3 | HCV GT4 | HCV GT5 | HCV GT6 | Total
Number analyzed (Participants) | 78 | 47 | 61 | 56 | 18 | 22 | 282
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.9 (12.6) | 52.7 (11.9) | 48.4 (10.1) | 46.4 (13.0) | 57.4 (12.4) | 53.3 (11.0) | 49.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 24 | 27 | 23 | 11 | 6 | 126
  Male | 43 | 23 | 34 | 33 | 7 | 16 | 156
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 0 | 1 | 22 | 29
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 1 | 0 | 0 | 4
  Black or African American | 4 | 0 | 1 | 8 | 9 | 0 | 22
  White | 69 | 44 | 57 | 47 | 4 | 0 | 221
  More than one race | 1 | 0 | 1 | 0 | 4 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Completing Study Therapy (SVR12)
Description: Plasma levels of hepatitis C virus (HCV) ribonucleic acid (RNA) were measured using the Roche COBAS® AmpliPrep/COBAS® TaqMan® HCV Test, v2.0 on blood samples drawn from participants. SVR12 is the absence of detectable RNA of the hepatitis C virus, (<lower limit of quantification [LLOQ] of 15 IU/mL) for at least 12 weeks after completing treatment.
Time Frame: 12 weeks after completing study therapy (Week 24)
Population: All participants who were assigned to treatment, and received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HCV GT1 | HCV GT2 | HCV GT3 | HCV GT4 | HCV GT5 | HCV GT6
Number analyzed (Participants) | 78 | 47 | 61 | 56 | 18 | 22
Percentage of participants | 92.3 [84.0 to 97.1] | 91.5 [79.6 to 97.6] | 73.8 [60.9 to 84.2] | 98.2 [90.4 to 100.0] | 100.0 [81.5 to 100.0] | 90.9 [70.8 to 98.9]

2. Primary Outcome: Percentage of Participants Experiencing an Adverse Event (AE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example ), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change infrequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to Week 14
Population: All participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | HCV GT1 | HCV GT2 | HCV GT3 | HCV GT4 | HCV GT5 | HCV GT6
Number analyzed (Participants) | 78 | 47 | 61 | 56 | 18 | 22
Percentage of participants | 60.3 | 61.7 | 57.4 | 55.4 | 77.8 | 77.3

3. Primary Outcome: Percentage of Participants Experiencing an AE of Clinical Importance (ECI)
Description: Adverse events of clinical importance, excluding overdoses include, but is not limited to, significant changes in alanine aminotransferase, aspartate aminotransferase, blood creatinine, glomerular filtration rate or hepatitis B reactivation.
Time Frame: Up to Week 14
Population: All participants who received at least one dose of study treatment
Measure: Number; unit: Percentage of participants
Arm/Group | HCV GT1 | HCV GT2 | HCV GT3 | HCV GT4 | HCV GT5 | HCV GT6
Number analyzed (Participants) | 78 | 47 | 61 | 56 | 18 | 22
Percentage of participants | 1.3 | 2.1 | 1.6 | 3.6 | 0 | 0

4. Primary Outcome: Percentage of Participants Experiencing a Serious Adverse Event (SAE)
Description: A serious adverse event (SAE) is any AE occurring at any dose or during any use of Sponsor's product that: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is an other important medical event; is a cancer; is associated with an overdose.
Time Frame: Up to Week 14
Population: All participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | HCV GT1 | HCV GT2 | HCV GT3 | HCV GT4 | HCV GT5 | HCV GT6
Number analyzed (Participants) | 78 | 47 | 61 | 56 | 18 | 22
Percentage of participants | 3.8 | 2.1 | 1.6 | 3.6 | 0 | 0

5. Primary Outcome: Percentage of Participants Experiencing a Drug-related AE
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example ), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change infrequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. A drug-related AE is determined by the investigator to be related to the use of the drug.
Time Frame: Up to Week 14
Population: All participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | HCV GT1 | HCV GT2 | HCV GT3 | HCV GT4 | HCV GT5 | HCV GT6
Number analyzed (Participants) | 78 | 47 | 61 | 56 | 18 | 22
Percentage of participants | 37.2 | 27.7 | 36.1 | 28.6 | 50.0 | 22.7

6. Primary Outcome: Percentage of Participants Experiencing a Drug-related SAE
Description: A SAE is any AE occurring at any dose or during any use of Sponsor's product that: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is an other important medical event; is a cancer; is associated with an overdose. A drug-related SAE is determined by the investigator to be related to the use of the drug.
Time Frame: Up to Week 14
Population: All participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | HCV GT1 | HCV GT2 | HCV GT3 | HCV GT4 | HCV GT5 | HCV GT6
Number analyzed (Participants) | 78 | 47 | 61 | 56 | 18 | 22
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Percentage of Participants Discontinuing Study Therapy Due to an AE
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example ), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change infrequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to Week 12
Population: All participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | HCV GT1 | HCV GT2 | HCV GT3 | HCV GT4 | HCV GT5 | HCV GT6
Number analyzed (Participants) | 78 | 47 | 61 | 56 | 18 | 22
Percentage of participants | 1.3 | 2.1 | 1.6 | 1.8 | 0 | 4.5

8. Secondary Outcome: Percentage of Participants With SVR 24 Weeks After Completing Study Therapy (SVR24)
Description: Plasma levels of HCV RNA) were measured using the Roche COBAS® AmpliPrep/COBAS® TaqMan® HCV Test, v2.0 on blood samples drawn from participants. SVR24 is the absence of detectable RNA of the hepatitis C virus (<LLOQ of 15 IU/mL), for at least 24 weeks after completing treatment.
Time Frame: 24 weeks after completing study therapy (Week 36)
Population: All participants who were assigned to treatment, and received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HCV GT1 | HCV GT2 | HCV GT3 | HCV GT4 | HCV GT5 | HCV GT6
Number analyzed (Participants) | 78 | 47 | 61 | 56 | 18 | 22
Percentage of participants | 89.7 [80.8 to 95.5] | 85.1 [71.7 to 93.8] | 72.1 [59.2 to 82.9] | 96.4 [87.7 to 99.6] | 100.0 [81.5 to 100.0] | 81.8 [59.7 to 94.8]

9. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure is the detection of HCV RNA among participants who do not discontinue study for non-treatment-related reasons, either due to on-treatment failure defined as either non-response where HCV RNA is detected at end of treatment without HCV RNA <LLOQ having been achieved while on treatment; rebound defined as >1 log10 IU/mL increase in HCV RNA from nadir while on treatment and confirmed from a separate blood draw within 2 weeks; or virologic breakthrough which is confirmed HCV RNA ≥LLOQ (target detected, quantifiable [TD(q)]) after being <LLOQ previously while on treatment. Confirmation is defined as an HCV RNA ≥LLOQ from a separate blood draw repeated within 2 weeks; or relapse post-treatment. where there is a confirmed HCV RNA ≥LLOQ [TD(q)] following end of all study therapy, after becoming undetectable (target not detected [TND]) at end of treatment. Confirmation is defined as an HCV RNA ≥LLOQ from a separate blood draw repeated within 2 weeks.
Time Frame: Up to Week 24
Population: Participants who followed the protocol sufficiently to allow the analysis of the results. Participants who deviated substantially from the protocol were excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | HCV GT1 | HCV GT2 | HCV GT3 | HCV GT4 | HCV GT5 | HCV GT6
Number analyzed (Participants) | 78 | 47 | 61 | 56 | 18 | 22
Percentage of participants | 3.8 | 2.1 | 23.0 | 0 | 0 | 13.6

ADVERSE EVENTS:
Time Frame: Up to Week 14
Description: All participants who received at least one dose of study treatment.
Arm/Group | HCV GT1 | HCV GT2 | HCV GT3 | HCV GT4 | HCV GT5 | HCV GT6
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/47 | 0/61 | 0/56 | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 3/78 | 1/47 | 1/61 | 2/56 | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 28/78 | 20/47 | 30/61 | 22/56 | 14/18 | 10/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCV GT1 (N=78) | HCV GT2 (N=47) | HCV GT3 (N=61) | HCV GT4 (N=56) | HCV GT5 (N=18) | HCV GT6 (N=22)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ammonia increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCV GT1 (N=78) | HCV GT2 (N=47) | HCV GT3 (N=61) | HCV GT4 (N=56) | HCV GT5 (N=18) | HCV GT6 (N=22)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (9) | 1 (1) | 4 (5) | 5 (6) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Asthenia (General disorders) | 5 (5) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 14 (16) | 5 (5) | 5 (5) | 4 (4) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 1 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (4) | 2 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 4 (4) | 3 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (11) | 5 (6) | 10 (13) | 8 (10) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT02956629/Prot_SAP_000.pdf